CLINICAL TRIAL: NCT06472895
Title: A Study of AK112 Monotherapy in Advanced/Metastatic Renal Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, MD, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK112-001-II-RCC
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Renal Cell Carcinoma
Keywords: RCC，immunotherapy，AK112，first-line treatment
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Subjects will receive AK112 (RP2D, administered intravenously，Q3W)
  Interventions: Drug: AK112 monotherapy

INTERVENTIONS:
Drug: AK112 monotherapy — A novel PD-1/VEGF bispecific antibody; RP2D intravenously (IV)，Q3W

SUMMARY:
This is an open-label, single arm , Ib/II phase trial to evaluate the efficacy and safety of AK112（ivonescimab）monotherapy as first-line treatment for favourable risk advanced/metastatic renal cell carcinoma (a/m RCC).

Subjects will receive AK112 until disease progression, unacceptable toxic effects, death，a decision by the physician or patient to withdraw from the trial，or AK112 exposure over 2 years.

The study set dose exploration stage and dose expansion stage respectively. Firstly, include a few subjects for observation in dose exploration stage, and select appropriate dose to enter expansion, then continue to include more subjects to further assessment.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent/assent for the trial.
* Be ≥18 and ≤ 75 years of age on day of signing informed consent, no matter male or female.
* IMDC favourable risk（IMDC score 0）.
* ECOG PS 0-1.
* Have estimated life expectancy of at least 3 months.
* Have histologically or cytologically confirmed diagnosis of RCC with mainly clear cell carcinoma component.
* Have received no prior systemic therapy for advanced RCC，Including but not limited to Immunotherapy, target therapy, chemotherapy, biological therapy, etc.

Note: Prior neoadjuvant/adjuvant therapies are acceptable if disease progression occurred > 6 months after last dosage of neoadjuvant/adjuvant treatment.

* Have measurable disease per RECIST v1.1 .
* Adequate organ function.
* Contraception from entering the trial，until 120 days after the last administration of the investigational drug.
* Willing to comply with the scheduled visits, treatment plans, and other requirements of the trial.

Exclusion Criteria:

* non-clear cell renal cell carcinoma，nccRCC（e.g. chromophobe, papillary)
* Has active autoimmune disease that might deteriorate when receiving an immunostimulatory agents. Subjects with diabetes type I, vitiligo, psoriasis, hypo-or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
* Has a known additional malignancy that has progressed or has required active treatment in the last 5 years.

Note: Subjects with basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or carcinoma in situ are not excluded.

* Eligible for surgery.
* History of severe bleeding or coagulation disorders.
* History of abdominal fistula or gastrointestinal perforation related to anti VEGF therapy.
* Has previously received systemic therapy.
* Has newly diagnosed brain metastases or known symptomatic brain metastases requiring steroids.
* Had major surgery 4 weeks prior to receiving first dose of trial treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 14 days prior to receiving first dose of trial treatment.
* Has an active tuberculosis and syphilitic infection.
* Has a known history of Human Immunodeficiency Virus (HIV) infection (HIV antibodies).
* Has known active Hepatitis B (e.g., Hepatitis B surface antigen [HBsAg] reactive and HBV-DNA>2000 IU/ml) or Hepatitis C virus (e.g., HCV RNA [qualitative] is detected).
* Has been pregnant or breastfeeding.
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-20 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
ORR per RECIST v1.1 assessed by investigators | Up to 2 years
  ORR is the proportion of subjects with complete response(CR) and partial response(PR) , based on RECIST v1.1

SECONDARY OUTCOMES:
DCR per RECIST v1.1 as assessed by investigators | Up to 2 years
  DCR is the proportion of subjects with complete response(CR), partial response(PR) and stable disease (SD) based on RECIST v1.1
Duration of response (DOR) | Up to 2 years
  Duration of response (DOR) assessed according to RECIST v1.1
Progression-free survival (PFS) | 3 years
  PFS is defined as the time from the the start of treatment till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the investigator or death due to any cause (whichever occurs first).
Overall survival (OS) | 4 years
  OS is the time from the first use of a therapeutic drug to death from any cause
Treatment-related adverse events | 3 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0, also types and degree